CLINICAL TRIAL: NCT03119155
Title: Improvement on Diagnosis of Fetal Congenital Heart Disease Based on Multi-center Collaboration in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, He Yihua,MD, Director of Department of Ultrosound, Beijing Anzhen Hospital
Other Study IDs: FCHD-CHINA01
Record Dates: First submitted 2017-04-13; First posted 2017-04-18 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Congenital Heart Disease; Echocardiography; Diagnosis
Keywords: Congenital Heart Disease; Echocardiography; Diagnosis
MeSH Terms: conditions — Heart Defects, Congenital; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to improve the diagnosis level of fetal congenital heart disease by the multi-center collaboration in China.

DETAILED DESCRIPTION:
Our center has constructed multi-center collaborative network in 2013, so far which contains more than 170 maternal and child health care hospitals throughout the whole of China. This is a multi-center-based study to improve the integral diagnostic level of fetal congenital heart diseases by fetal echocardiography. Sixty pregnant cases (18-45 years) whose fetuses with heart abnormalities will be recruited in a successive manner from every center every year. Cases are gravidas with fetal congenital heart disease diagnosed by echocardiography in 16th-24th of gestational weeks. Every center will upload the echocardiography materials and the diagnostic reports so that another two experienced echocardiography physicians confirm the diagnosis based on these materials in a double-blinded method. In addition, the golden standard of congenital heart disease depends on the autopsy, heart and vascular casting after abortion and operation after birth. The investigators will provide the report about the rate of missed diagnosis and misdiagnosis and the periodical training on fetal echocardiography for every center every half an year. Only gravidas who are willing to have complete pregnancy checks and finally delivery or abortion in the hospital are interviewed are eligible for the study. Study participants will be asked for their informed consent.

ELIGIBILITY:
Inclusion Criteria:

* 1.Gravida with singleton pregnancy with congenital heart disease taking fetal echocardiography in 16th-24nd of gestational weeks.
* 2.Complete pregnancy check in Beijing Anzhen Hospital and the hospitals contained in our multi-center network collaboration, and finally delivery or abortion in these hospitals.
* 3.Willing to cooperate with our study.

Exclusion Criteria:

* 1. Pregnant women with serious pregnancy complications and suffering from mental illness.
* 2.Pregnant women not willing to cooperate

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Gravidas with singleton pregnancy with congenital heart disease
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
the rate of missed diagnosis and misdiagnosis | From Jan 2018 to Dec 2020
  We will report the primary outcome every year, and compare the change trend of diagnostic level of fetal congenital heart disease

SECONDARY OUTCOMES:
The prognosis of different type of fetal congenital heart disease with 1 year after birth | From Jan 2018 to Dec 2021
  We will get the abortion rate of different types of fetal congenital heart disease and operation rate within 1 year after birth.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijng Anzhen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided